CLINICAL TRIAL: NCT04734132
Title: Effects of Moringa Oleifera Leaves on Glycemia, Lipemia and Inflammatory Profile. Nutritional Intervention Study in Prediabetic Patients
Brief Title: Effects of Moringa Oleifera Leaves on Glycemia, Lipemia and Inflammatory Profile in Prediabetic Patients
Acronym: NUTRIMOL-DB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Esther Nova Rebato, Principal Investigator, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AGL2017-86044-C2-1-R
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: PreDiabetes
Keywords: Moringa oleifera; functional food; anti-hyperglycemic effect; prevention; anti-inflammatory; microbiota; lipid metabolism
MeSH Terms: conditions — Prediabetic State | interventions — flocculant protein MO 2.1, Moringa oleifera

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, parallel group, placebo-controlled dietary intervention in prediabetic subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One member of the research team was in charge of product preparation and delivery to the participants following the randomization list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa (Experimental): Six Moringa oleifera capsules (400 mg dry leaf powder /capsule) consumed daily during 12 weeks. Two capsules consumed with each of the three main meals.
  Interventions: Dietary Supplement: Moringa
- Placebo (Placebo Comparator): Six placebo capsules containing microcrystalline cellulose consumed daily during 12 weeks. Two capsules consumed with each of the three main meals.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Moringa — Leaves of Moringa oleifera from an organic Iberian peninsula cultivar. A single lot was prepared from the same crop. Leaves were dried and ground and encapsulated as a organic dietary supplement. No other changes in diet or physical activity were included although a general healthy lifestyle pattern was recommended.
  Arms: Moringa
Dietary Supplement: Placebo — Placebo capsules were indistinguishable from the experimental capsules in material and color (opaque white). Same number of capsules were consumed as in the experimental arm and no other changes in diet or physical activity were included although a general healthy lifestyle pattern was recommended.
  Arms: Placebo

SUMMARY:
Moringa oleifera (MO) is a traditional food in tropical and subtropical areas and has attained a growing interest for its medicinal properties. It's a nutrient-rich vegetable, high in protein and polyphenol content. The MO dry leaves and leaf extracts have been shown to exert numerous in vitro activities and in vivo effects, including the hypoglycemic effect. Thus, MO could be an alternative to prevent or treat diabetes. Studies in humans, however, are still limited. This proposal aims to study the efficacy of Moringa oleifera to improve the control of glycaemia in subjects with prediabetes. A 3-month dietary intervention with MO dry leave capsules will be performed and compared to placebo.

DETAILED DESCRIPTION:
The tree Moringa oleifera (MO) is a traditional medicinal plant in tropical and subtropical areas, also consumed as food, which is currently expanding worldwide as a protein-rich leafy vegetable and for the medicinal value of its phytochemicals, in particular its glucosinolates. Specifically, MO dry leaves and leaf extracts have been shown to exert numerous in vitro activities and in vivo effects, including the hypoglycemic effect. Thus, MO could be an alternative to prevent or treat diabetes. In this sense, in vitro and preclinical experiments have shown that MO could potentially reverse some of the pathophysiological manifestation of diabetes and its comorbidities, such as hepatic fat accumulation and insulin resistance, oxidative stress, inflammation and peripheral hyperglycemia. Studies in humans, however, are still limited. This proposal aims to study the efficacy of Moringa oleifera to improve the control of glycaemia in subjects with prediabetes. A 3-month dietary intervention with MO dry leave capsules will be performed and compared to placebo. This will be a double-blind, randomized, placebo controlled, parallel group intervention study. Subjects will randomly consume either 6 capsules of dry MO leaves (400 mg dry leaf powder /capsule) or 6 placebo capsules per day during 3 months. The study subjects will provide samples for outcome measurements at three different time points: basal, 6 weeks and 12 weeks of supplementation. Glycaemia and plasma inflammatory and metabolic markers will be measured, as well as the gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetes: HbA1c between 5.7-6.4 % or fasting blood glucose between 100 - 125 mg/dl or impaired glucose tolerance (> 140 mg/dl and < 200 mg/dl two hours post oral challenge).
* No pharmacological treatment prescribed for glycemia control.

Exclusion Criteria:

* Diabetes Mellitus
* Impaired renal function: < 60% Glomerular filtration
* Uncontrolled high blood pressure
* Previous cardiovascular events or coronary disease
* Autoimmune disease
* HIV
* Severe gastrointestinal disease
* Cancer
* Psychiatric illness
* Elevated liver enzymes (x2 normal range)
* Alcohol abuse (higher than 14 and 21 doses/week for women and men, respectively)
* Morbid obesity (BMI>35kg/m2)
* Pregnancy
* Pharmacological treatments that interfere with glucose control.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | 12 weeks
  Measured in serum samples from fasting blood withdrawn in a Sodium Fluoride vacutainer tube
Glycated hemoglobin (HbA1C) | 12 weeks
  Measured in fasting serum

SECONDARY OUTCOMES:
Conversion rate from prediabetes to normal | 12 weeks
  Number of subjects in each arm that convert from prediabetic to normal glycemia

OTHER OUTCOMES:
Total serum cholesterol concentration and lipoprotein-cholesterol concentrations | 12 weeks
  Serum lipid profile
Concentration of inflammatory markers | 12 weeks
  C-reactive protein, interleukin (IL)-1beta, IL-6, Tumour necrosis factor-alpha, Macrophage chemoattractant protein-1
Concentration of metabolic hormones | 12 weeks
  Insulin, Glucagon like peptide-1, Peptide YY, leptin, adiponectin, ghrelin,
Antioxidant capacity | 12 weeks
  Total antioxidant capacity of the lipid soluble fraction of plasma by chemiluminescent method (Photochem)
Microbiota composition | 12 weeks
  Quantitative analysis of main representative bacteria groups of gut microbiota by quantitative polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Esther NOVA, PhD, Principal Investigator — National Research Council of Spain
Locations (1):
- Institute of Food Science and Technology and Nutrition (ICTAN)-CSIC, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Although a specific plan has not been conceived yet, sharing research data is a good practice that the investigators would pursue at due time.

REFERENCES:
- [Background] Nova E, Redondo-Useros N, Martinez-Garcia RM, Gomez-Martinez S, Diaz-Prieto LE, Marcos A. Potential of Moringa oleifera to Improve Glucose Control for the Prevention of Diabetes and Related Metabolic Alterations: A Systematic Review of Animal and Human Studies. Nutrients. 2020 Jul 10;12(7):2050. doi: 10.3390/nu12072050. PMID 32664295
- [Background] Vargas-Sanchez K, Garay-Jaramillo E, Gonzalez-Reyes RE. Effects of Moringa oleifera on Glycaemia and Insulin Levels: A Review of Animal and Human Studies. Nutrients. 2019 Dec 2;11(12):2907. doi: 10.3390/nu11122907. PMID 31810205